CLINICAL TRIAL: NCT05776225
Title: Pulmonary Hypertension Screening in Patients With Interstitial Lung Disease for Earlier Detection (PHINDER)
Brief Title: Pulmonary Hypertension Screening in Patients With Interstitial Lung Disease for Earlier Detection
Acronym: PHINDER
Status: Recruiting | Type: Observational
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: GMS-PH-001
Record Dates: First submitted 2023-03-01; First posted 2023-03-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Interstitial Lung Disease; Pulmonary Hypertension
Keywords: ILD; PH; PH-ILD
MeSH Terms: conditions — Lung Diseases, Interstitial; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental study arm: All enrolled patients in this single arm study will receive a RHC.
  Interventions: Procedure: Right heart catheterization (RHC)

INTERVENTIONS:
Procedure: Right heart catheterization (RHC) — RHC to evaluate pulmonary hemodynamics

SUMMARY:
Study GMS-PH-001 is a multicenter, open-label, non-randomized study to prospectively evaluate screening strategies of pulmonary hypertension (PH) in patients with interstitial lung disease (ILD).

DETAILED DESCRIPTION:
In this study, subjects will undergo a broad range of clinical assessments that are potentially associated with PH. Study data will be used to identify and weigh specific clinical parameters based on their prognostic significance for right heart catheterization (RHC)-confirmed PH. There is no study drug under investigation in this study. The study consists of 2 study visits: a Screening Visit and Study Visit 1.

Clinical assessments include pulmonary function tests (PFTs); high resolution computed tomography (HRCT); physical examination; 6-Minute Walk Test; blood draw for clinical laboratory parameters, plasma brain natriuretic peptide (BNP) concentration and plasma N-terminal pro-BNP (NT-proBNP) concentration; echocardiography; University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ); King's Brief Interstitial Lung Disease Questionnaire (K-BILD); 36-Item Short Form Survey (SF-36); Pulmonary Hypertension Functional Classification Self Report (PH-FC-SR); Investigator's Suspicion of PH Questionnaire; adverse event (AE) monitoring; and RHC.

As the primary objective of this study is to collect a broad range of clinical parameters in patients with ILD, it is expected that numerous exploratory and post-hoc analyses will be performed to identify and weigh specific parameters based on their prognostic significance for PH in this patient population with the goal of developing a screening algorithm for PH in patients with ILD.

ELIGIBILITY:
Inclusion Criteria

1. Patient gives voluntary written informed consent to participate in the study and are capable of reading and understanding questionnaires or forms in English or Spanish.
2. Patients with a diagnosis of ILD based on computed tomography imaging, including:

   1. Idiopathic interstitial pneumonia, including idiopathic pulmonary fibrosis
   2. Connective tissue disease-associated ILD with forced vital capacity (FVC) <70%
   3. Hypersensitivity pneumonitis
   4. Scleroderma-related ILD
   5. Autoimmune ILD
   6. Nonspecific interstitial pneumonia
   7. Occupational lung disease
   8. Combined pulmonary fibrosis and emphysema with mild emphysema on lung imaging as determined by the Investigator
3. Patients must have at least 2 signs or symptoms suggestive of PH, as specified by the study protocol.

Exclusion Criteria

1. Prior RHC with mPAP >20 mmHg.
2. Currently on a Food and Drug Administration (FDA)-approved pulmonary arterial hypertension (PAH) medication for the treatment of PAH.
3. Diagnosed with chronic obstructive pulmonary disease (CPFE with mild emphysema notwithstanding).
4. Uncontrolled or untreated moderate to severe sleep apnea as determined by the patient's physician.
5. Pulmonary embolism within the past 3 months.
6. History of ischemic heart disease or left-sided myocardial dysfunction within 12 months of Screening, defined as left ventricular ejection fraction <40% or pulmonary capillary wedge pressure >15 mmHg.
7. Any other clinical features that, in the opinion of the Investigator, might adversely affect interpretation of study data or study safety, or make the patient unsuitable for RHC or HRCT (e.g., pregnancy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PH-ILD being treated in any setting, including academic, community, etc.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with PH as indicated by RHC | Through study completion, approximately 3 weeks.
  Mean pulmonary artery pressure (mPAP) >20 mmHg with pulmonary artery wedge pressure (PAWP) ≤15 mmHg and pulmonary vascular resistance (PVR) >2 WU.

SECONDARY OUTCOMES:
Percentage of patients with severe PH as indicated by RHC | Through study completion, approximately 3 weeks.
  mPAP >20 mmHg with PAWP ≤15 mmHg and PVR >5 WU.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Pulmonary Associates, Phoenix, Arizona
  - Hartford Hospital, Hartford, Connecticut
  - Lakeland Regional Health, Lakeland, Florida
  - NCH Healthcare System, Naples, Florida
  - University of South Florida Health, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Healthcare, Austell, Georgia
  - Loyola University Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - NorthShore University Health System, Glenview, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - LSU Health Sciences Center New Orleans, New Orleans, Louisiana
  - University of Michigan Int Med Pulmonary and Critical Care, Ann Arbor, Michigan
  - Mclaren Greater Lansing, Okemos, Michigan
  - Blessing Health Hannibal, Hannibal, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Pulmonix, LLC, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Legacy Health, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - AnMed Health Pulmonary and Sleep Medicine, Anderson, South Carolina
  - Prisma Health, Columbia, South Carolina
  - StatCare Pulmonary Consultants, Knoxville, Tennessee
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Healthcare, Murray, Utah
  - University of Utah Health, Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - Providence Medical Research Center, Spokane, Washington
  - Marshall Health, Huntington, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Kulkarni T, Zisman DA, Shlobin OA, Kiely DG, DerSarkissian M, Shen E, Maher KM, Broderick M, Scholand MB. Study Design and Rationale for the PHINDER Study: Pulmonary Hypertension Screening in Patients with Interstitial Lung Disease for Earlier Detection. Pulm Ther. 2025 Sep;11(3):491-501. doi: 10.1007/s41030-025-00307-0. Epub 2025 Jul 25. PMID 40711711